CLINICAL TRIAL: NCT02448706
Title: Characterizing Variability in Hearing Aid Outcomes Among Older Adults
Brief Title: Variability In Hearing Aid Outcomes In Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Pamela Souza, Professor School of Communication, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1R01DC012289-01 (NIH); 1R01DC012289-01 (NIH)
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Hearing Loss; Presbycusis
Keywords: hearing aid
MeSH Terms: conditions — Hearing Loss; Presbycusis | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hearing Aid Fitting Order A (Active Comparator): High level of signal manipulation for 6 weeks, followed by a low level of signal manipulation for 6 weeks.
  Interventions: Device: Hearing Aid Fitting A; Device: Hearing Aid Fitting B
- Hearing Aid Fitting Order B (Active Comparator): Low level of signal manipulation for 6 weeks, followed by a low level of signal manipulation for 6 weeks.
  Interventions: Device: Hearing Aid Fitting A; Device: Hearing Aid Fitting B

INTERVENTIONS:
Device: Hearing Aid Fitting A
  Other Names: Hearing Aid
Device: Hearing Aid Fitting B

SUMMARY:
The goal of this project is to find out if the way a hearing aid processes a sound signal should be determined in part by an individual's cognitive characteristics. We anticipate that the outcome of this work will be a battery of assessments that will guide hearing aid processing for older patients with hearing loss.

DETAILED DESCRIPTION:
Response to hearing aids is highly variable, with some individuals reporting much more benefit than others. Preliminary work by our laboratory and others suggests that patient factors-including cognition-may contribute to differences in how individuals respond to altered speech cues, such as those alterations introduced by hearing aid processing. The long-term goal of this work is to improve hearing aid outcomes by optimizing hearing aid processing for each individual.

ELIGIBILITY:
Inclusion Criteria:

* Sensorineural Hearing loss with pure-tone thresholds 25-70 dB HL at octave frequencies between 250 and 4000 Hz, 4 frequency PTA of ≥ 30 dB HL
* Non hearing aided wearer within the previous year
* Participants will be in good health (self-report)
* Normal or corrected to normal vision(≤20/50)

Exclusion Criteria:

* Conductive, or asymmetric hearing loss
* Hearing loss exceeding the limits that can be successfully aided with hearing aids (i.e., profound hearing loss)
* Hearing loss remediated with a cochlear implant (cannot wear hearing aids)
* Significant history of otologic or neurologic disorders
* Non English speaking participants
* Score of 23 or below on Mini-Mental Status Exam (MMSE)
* Score of 22 or below on Montreal Cognitive Assessment (MoCA)
* Any clinically significant unstable or progressive medical condition
* Any condition which, in the opinion of the investigator, places the participant at unacceptable risk if he or she were to participate in the study.
* Participants will be divided into low and high working groups based upon the results of their Lunner working memory reading span test. Once either high or low working memory group is filled (approximately 25 participants) we will selectively enroll participants to fill the other category.

Min Age: 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela E Souza, PhD, Principal Investigator — Northwestern University; Kathryn H Arehart, PhD, Principal Investigator — University of Colorado at Boulder
Locations (1):
- University of Colorado at Boulder, Boulder, Colorado, United States

REFERENCES:
- [Derived] Anderson M, Rallapalli V, Schoof T, Souza P, Arehart K. The use of self-report measures to examine changes in perception in response to fittings using different signal processing parameters. Int J Audiol. 2018 Nov;57(11):809-815. doi: 10.1080/14992027.2018.1490035. Epub 2018 Jul 27. PMID 30052097

RESULTS

PARTICIPANT FLOW:
Groups:
- Hearing Aid Fitting Order A: High level of signal manipulation (5 weeks), then low level of signal manipulation (5 weeks)
- Hearing Aid Fitting Order B: Low level of signal manipulation (5 weeks), then high level of signal manipulation (5 weeks)
Period: Overall Study
Arm/Group | Hearing Aid Fitting Order A | Hearing Aid Fitting Order B
Started | 25 | 24
Withdrew for Personal Reasons | 1 | 1
Completed Baseline Testing | 24 | 23
Completed | 20 | 20
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants received the same baseline measures, regardless of the hearing aid fitting order to which they were randomized
Arm/Group | All Study Participants
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 38
Age, Continuous [Mean (Full Range); unit: years] | 72 [54 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 47
Reading span task [Mean (Full Range); unit: percentage of correctly recalled words] — Participants view a series of sentences on a computer screen. For each sentence, participants are asked to make a judgment as to whether the sentence makes semantic sense (processing task). After a block of sentences, the participant is asked to recall either first of last words of the sentences (storage task). Final score is the percentage of correctly recalled words.
  percentage of correctly recalled words | 34 [11 to 56]

OUTCOME MEASURES:

1. Primary Outcome: Speech Intelligibility Score
Description: Participants listen to sentences in a background of noise and repeat the sentence heard. The outcome is percentage of correctly repeated words.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Groups:
- High Level of Signal Manipulation: Fit with hearing aids set to a high level of signal manipulation (6 weeks). Half of the participants completed this condition in the first 6 weeks of the trial, and half in the second 6 weeks of the trial.
- Low Level of Signal Manipulation: Fit with hearing aids set to a low level of signal manipulation (6 weeks). Half of the participants completed this condition in the first 6 weeks of the trial, and half in the second 6 weeks of the trial.
Arm/Group | High Level of Signal Manipulation | Low Level of Signal Manipulation
Number analyzed (Participants) | 40 | 40
percentage of correct responses | 69 (18) | 78 (15)

2. Secondary Outcome: Effectiveness of Aural Rehabilitation (EAR)
Description: The listener rates the extent to which hearing has improved with the hearing aid (0=least improved, 100=most improved).
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Hearing Aid Fitting A: High level of signal manipulation
  Hearing Aid Fitting A
- Hearing Aid Fitting B: Low level of signal manipulation
  Hearing Aid Fitting B
Arm/Group | Hearing Aid Fitting A | Hearing Aid Fitting B
Number analyzed (Participants) | 40 | 40
score on a scale | 60.0 (23.3) | 74.2 (21.0)

3. Secondary Outcome: Speech and Spatial Qualities of Hearing (SSQ) Questionnaire
Description: Listener rates her/his perceived ability. Each question describes a different situation, such as listening to one talker in quiet. Test is scored from 0 to 10, with 10 = best score.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hearing Aid Fitting A | Hearing Aid Fitting B
Number analyzed (Participants) | 40 | 40
score on a scale | 6.47 (1.4) | 6.95 (1.1)

4. Secondary Outcome: Adherence
Description: Average number of hours per day the hearing aid was worn.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Hearing Aid Fitting A | Hearing Aid Fitting B
Number analyzed (Participants) | 40 | 40
hours per day | 9 (3.7) | 9 (3.4)

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Hearing Aid Fitting A: High level of signal manipulation
- Hearing Aid Fitting B: Low level of signal manipulation
Arm/Group | Hearing Aid Fitting A | Hearing Aid Fitting B
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT02448706/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT02448706/ICF_001.pdf